CLINICAL TRIAL: NCT01346358
Title: Phase 1 Study of IMC-CS4, a Monoclonal Antibody Targeted to the CSF-1 Receptor (CSF-1R), In Subjects With Advanced Solid Tumors Refractory to Standard Therapy or for Which No Standard Therapy is Available
Brief Title: A Study of IMC-CS4 in Subjects With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 14311; CP24-1001 (Other: ImClone Systems); I5F-IE-JSCA (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-04-29; First posted 2011-05-03 (Estimated); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-05

CONDITIONS: Neoplasms
Keywords: Advanced Solid Tumors
MeSH Terms: conditions — Neoplasms | interventions — LY3022855

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IMC-CS4 Weight Based Dosing (Experimental): Participants received 2.5 mg/kg once weekly (QW), 0.3 mg/kg QW, 0.6 mg/kg QW, 1.25 mg/kg every two weeks (Q2W) and1.25 mg/kg QW of IMC CS4 by intravenous infusion in Part A.
  Interventions: Biological: IMC-CS4
- IMC-CS4 Non-Weight Based Dosing (Experimental): Participants received 100 mg QW, 100 mg QW on weeks 1, 2, 4 and 5 and 150 mg QW of IMC CS4 by intravenous infusion in Part B.
  Interventions: Biological: IMC-CS4

INTERVENTIONS:
Biological: IMC-CS4
  Other Names: LY3022855

SUMMARY:
A dose escalation study to establish the safety profile and characterize the pharmacokinetic profile of IMC-CS4 in the treatment of subjects with advanced solid tumors refractory to standard therapy or for which no standard therapy is available.

ELIGIBILITY:
Inclusion Criteria:

* Subject has histologic or cytologic confirmation of advanced solid tumors that is refractory to standard therapy or for which no standard therapy is available
* Subject has measurable or nonmeasurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
* Subject has resolution to grade ≤1 by NCI-CTCAE (Common Toxicity Criteria for Adverse Effects) Version 4.03 of all clinically significant toxic effects of prior treatment
* Subject has an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Subject has adequate hematologic, hepatic, renal, and coagulation function
* Subject has a life expectancy greater than 3 months
* Subject agrees to use adequate contraception during the study period and for 12 weeks after last dose of study therapy
* Subject must undergo mandatory biopsies, including one pretreatment and one post treatment tumor biopsy procedure

Exclusion Criteria:

* Subject has experienced acute pathologic fracture or spinal cord compression within 28 days prior to first dose of study therapy
* Subject has a known hypersensitivity to monoclonal antibodies or to agents of similar biologic composition as IMC-CS4.
* Subject has received treatment with any monoclonal antibodies within 4 weeks prior to first dose of study therapy
* Subject has undergone a major surgical procedure, open biopsy, radiofrequency ablation or has experienced a significant injury within 28 days prior to enrollment
* Subject has a concurrent active malignancy other than adequately treated nonmelanomatous skin cancer or in situ neoplasm
* Subject has an ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, active bleeding or any other serious uncontrolled medical disorder
* Subject has known or suspected primary brain or leptomeningeal metastases
* Subject has leukemia or lymphoma
* Subject is know to have active tuberculosis, leishmaniasis, or listeriosis
* Subjects with known history, or clinical or laboratory evidence of liver disease
* Subject has a known active hepatitis B or C infection, Human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome (AIDS)
* Subject if female, is pregnant or breastfeeding
* Subject has received an organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2011-06-15 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (6):
- United States (6):
  - The Angeles Clinic & Research Institute, Los Angeles, California
  - Univ of California San Francisco, San Francisco, California
  - Emory University, Atlanta, Georgia
  - Columbia University College of Phys & Surgeons, New York, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Ohio State University Medical Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dowlati A, Harvey RD, Carvajal RD, Hamid O, Klempner SJ, Kauh JSW, Peterson DA, Yu D, Chapman SC, Szpurka AM, Carlsen M, Quinlan T, Wesolowski R. LY3022855, an anti-colony stimulating factor-1 receptor (CSF-1R) monoclonal antibody, in patients with advanced solid tumors refractory to standard therapy: phase 1 dose-escalation trial. Invest New Drugs. 2021 Aug;39(4):1057-1071. doi: 10.1007/s10637-021-01084-8. Epub 2021 Feb 23. PMID 33624233

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Completers included participants who died from any cause or disease progression and participants who were alive and on study (either on study treatment or in long term follow-up) at study conclusion.
Groups:
- Cohort 1 (2.5 Milligram Per Kilogram (mg/kg) QW): Participants received 2.5 milligram per kilogram (mg/kg) of IMC-CS4 once weekly (QW) by intravenous infusion.
- Cohort 2 (0.3 mg/kg QW): Participants received 0.3 mg/kg of IMC-CS4 once weekly by intravenous infusion.
- Cohort 3 (0.6 mg/kg QW): Participants received 0.6 mg/kg of IMC-CS4 once weekly by intravenous infusion.
- Cohort 4 (1.25 mg/kg Q2W): Participants received 1.25 mg/kg of IMC-CS4 every two weeks (Q2W) by intravenous infusion.
- Cohort 4 Expanded (1.25 mg/kg Q2W): Participants received 1.25 mg/kg of IMC-CS4 every two weeks by intravenous infusion on weeks 1, 2, 4 and 5.
- Cohort 5 (1.25 mg/kg QW): Participants received 1.25 mg/kg of IMC-CS4 weekly once by intravenous infusion.
- Cohort 6a (100 mg QW): Participants received 100 mg of IMC-CS4 weekly once by intravenous infusion.
- Cohort 6a Expanded (100 mg QW): Participants received 100 mg of IMC-CS4 weekly once by intravenous infusion on weeks 1, 2, 4 and 5.
- Cohort 7a (150 mg QW): Participants received 150 mg of IMC-CS4 weekly once by intravenous infusion.
Period: Overall Study
Arm/Group | Cohort 1 (2.5 Milligram Per Kilogram (mg/kg) QW) | Cohort 2 (0.3 mg/kg QW) | Cohort 3 (0.6 mg/kg QW) | Cohort 4 (1.25 mg/kg Q2W) | Cohort 4 Expanded (1.25 mg/kg Q2W) | Cohort 5 (1.25 mg/kg QW) | Cohort 6a (100 mg QW) | Cohort 6a Expanded (100 mg QW) | Cohort 7a (150 mg QW)
Started | 6 | 4 | 3 | 6 | 5 | 5 | 3 | 11 | 9
Completed | 4 | 3 | 2 | 5 | 4 | 3 | 2 | 7 | 6
Not Completed | 2 | 1 | 1 | 1 | 1 | 2 | 1 | 4 | 3
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 1 | 0 | 2 | 1 | 1 | 1
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Not completed — Non-Compliance | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Groups:
- Cohort 1 (2.5 Milligram Per Kilogram (mg/kg) QW): Participants received 2.5 milligram per kilogram (mg/kg) of IMC-CS4 once weekly by intravenous infusion.
- Cohort 4 (1.25 mg/kg Q2W): Participants received 1.25 mg/kg of IMC-CS4 every two weeks by intravenous infusion.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (2.5 Milligram Per Kilogram (mg/kg) QW) | Cohort 2 (0.3 mg/kg QW) | Cohort 3 (0.6 mg/kg QW) | Cohort 4 (1.25 mg/kg Q2W) | Cohort 4 Expanded (1.25 mg/kg Q2W) | Cohort 5 (1.25 mg/kg QW) | Cohort 6a (100 mg QW) | Cohort 6a Expanded (100 mg QW) | Cohort 7a (150 mg QW) | Total
Number analyzed (Participants) | 6 | 4 | 3 | 6 | 5 | 5 | 3 | 11 | 9 | 52
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.3 (6.22) | 63.3 (1.71) | 65.0 (4.58) | 63.5 (12.57) | 60.8 (13.99) | 51.6 (12.62) | 54.0 (10.15) | 55.5 (12.26) | 59.1 (8.58) | 58.6 (10.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 2 | 1 | 4 | 2 | 2 | 7 | 3 | 25
  Male | 3 | 3 | 1 | 5 | 1 | 3 | 1 | 4 | 6 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 3
  Not Hispanic or Latino | 6 | 4 | 3 | 5 | 5 | 5 | 3 | 9 | 9 | 49
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 3 | 7
  White | 4 | 3 | 3 | 5 | 5 | 4 | 3 | 7 | 4 | 38
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 4 | 3 | 6 | 5 | 5 | 3 | 11 | 9 | 52

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK) - Maximum Concentration (Cmax) of IMC-CS4
Description: Pharmacokinetics (PK) - Maximum concentration (Cmax) of IMC-CS4.
Time Frame: Predose, 1, 2, 4 and 8 hours post dose of Cycle 1 Day 1, Cycle 1 Day 15, Cycle 1 Day 22 and Cycle 3 Day 1
Population: All enrolled participants who received at least one dose of study drug and have evaluable PK data for Cmax.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram/milliliters (µg/mL)
Groups:
- 2.5 mg/kg of IMC-CS4 QW: Participants received 2.5 milligram per kilogram (mg/kg) of IMC-CS4 once weekly by intravenous infusion.
- 0.3 mg/kg of IMC-CS4 QW: Participants received 0.3 mg/kg of IMC-CS4 once weekly by intravenous infusion.
- 0.6 mg/kg of IMC-CS4 QW: Participants received 0.6 mg/kg of IMC-CS4 once weekly by intravenous infusion.
- 1.25 mg/kg of IMC-CS4 QW; 1.25 mg/kg of IMC-CS4 Q2W: Participants received 1.25 mg/kg of IMC-CS4 every two weeks by intravenous infusion.
- 100 mg of IMC-CS4 QW: Participants received 100 mg of IMC-CS4 weekly once by intravenous infusion.
- 150 mg of IMC-CS4 QW: Participants received 150 mg of IMC-CS4 weekly once by intravenous infusion.
Arm/Group | 2.5 mg/kg of IMC-CS4 QW | 0.3 mg/kg of IMC-CS4 QW | 0.6 mg/kg of IMC-CS4 QW | 1.25 mg/kg of IMC-CS4 QW | 1.25 mg/kg of IMC-CS4 Q2W | 100 mg of IMC-CS4 QW | 150 mg of IMC-CS4 QW
Number analyzed (Participants) | 6 | 4 | 3 | 5 | 10 | 14 | 8
Microgram/milliliters (µg/mL)
  Cycle 1 Day 1 | 69.2 (13) | 6.83 (32) | 13.5 (33) | 26.0 (14) | 31.2 (24) | 32.2 (25) | 42.9 (20)
  Cycle 1 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 10 | 0 | 0
  Cycle 1 Day 15 |  |  |  |  | 30.0 (25) |  |
  Cycle 1 Day 22: number analyzed (Participants) | 4 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 1 Day 22 | 92.7 (23) |  |  |  |  |  |
  Cycle 3 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 5 | 1
  Cycle 3 Day 1 |  |  |  |  |  | 42.8 (59) | NA (NA) — Not analyzed due to insufficient number of participants.

2. Primary Outcome: Pharmacokinetics - Minimum Concentration (Cmin) of IMC-CS4
Description: Pharmacokinetics - Minimum concentration (Cmin) of IMC-CS4.
Time Frame: Predose, 1, 2, 4 and 8 hours post dose of Cycle 1 Day 1, Cycle 1 Day 15, Cycle 1 Day 22 and Cycle 3 Day 1
Population: All enrolled participants who received at least one dose of study drug and have evaluable PK data for Cmin.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | 2.5 mg/kg of IMC-CS4 QW | 0.3 mg/kg of IMC-CS4 QW | 0.6 mg/kg of IMC-CS4 QW | 1.25 mg/kg of IMC-CS4 QW | 1.25 mg/kg of IMC-CS4 Q2W | 100 mg of IMC-CS4 QW | 150 mg of IMC-CS4 QW
Number analyzed (Participants) | 6 | 0 | 0 | 2 | 5 | 9 | 8
µg/mL
  Cycle 1 Day 1 | 14.4 (34) |  |  | NA (NA) — Not analyzed due to insufficient number of participants. | 3.32 (11) | 3.77 (79) | 5.15 (81)
  Cycle 1 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 4 | 0 | 0
  Cycle 1 Day 15 |  |  |  |  | 3.35 (22) |  |
  Cycle 1 Day 22: number analyzed (Participants) | 6 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 1 Day 22 | 29.9 (36) |  |  |  |  |  |
  Cycle 3 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 4 | 1
  Cycle 3 Day 1 |  |  |  |  |  | 21.9 (86) | NA (NA) — Not analyzed due to insufficient number of participants.

3. Primary Outcome: Pharmacokinetics - Area Under the Curve (AUC) of IMC-CS4
Description: Pharmacokinetics - Area Under the Curve (AUC) of IMC-CS4.
Time Frame: Predose, 1, 2, 4 and 8 hours post dose of Cycle 1 Day 1, Cycle 1 Day 15, Cycle 1 Day 22 and Cycle 3 Day 1
Population: All enrolled participants who received at least one dose of study drug and have evaluable PK data for AUC.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours* microgram per mL (h*µg/mL)
Arm/Group | 2.5 mg/kg of IMC-CS4 QW | 0.3 mg/kg of IMC-CS4 QW | 0.6 mg/kg of IMC-CS4 QW | 1.25 mg/kg of IMC-CS4 QW | 1.25 mg/kg of IMC-CS4 Q2W | 100 mg of IMC-CS4 QW | 150 mg of IMC-CS4 QW
Number analyzed (Participants) | 6 | 3 | 3 | 5 | 10 | 14 | 8
Hours* microgram per mL (h*µg/mL)
  Cycle 1 Day 1 | 5020 (18) | 256 (14) | 492 (23) | 1810 (21) | 1550 (50) | 1780 (43) | 2810 (34)
  Cycle 1 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 9 | 0 | 0
  Cycle 1 Day 15 |  |  |  |  | 1700 (49) |  |
  Cycle 1 Day 22: number analyzed (Participants) | 3 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 1 Day 22 | 11300 (18) |  |  |  |  |  |
  Cycle 3 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 4 | 1
  Cycle 3 Day 1 |  |  |  |  |  | 4430 (80) | NA (NA) — Not analyzed due to insufficient number of participants.

4. Primary Outcome: Pharmacokinetics - Volume of Distribution at Steady State (Vss) of IMC-CS4
Description: Pharmacokinetics - Volume of distribution at steady state (Vss) of IMC-CS4.
Time Frame: Predose, 1, 2, 4 and 8 hours post dose of Cycle 1 Day 1, Cycle 1 Day 15, Cycle 1 Day 22 and Cycle 3 Day 1
Population: All enrolled participants who received at least one dose of study drug and have evaluable PK data for Vss.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters (L)
Arm/Group | 2.5 mg/kg of IMC-CS4 QW | 0.3 mg/kg of IMC-CS4 QW | 0.6 mg/kg of IMC-CS4 QW | 1.25 mg/kg of IMC-CS4 QW | 1.25 mg/kg of IMC-CS4 Q2W | 100 mg of IMC-CS4 QW | 150 mg of IMC-CS4 QW
Number analyzed (Participants) | 6 | 3 | 3 | 5 | 10 | 14 | 8
Liters (L)
  Cycle 1 Day 1 | 4.80 (40) | 4.61 (4) | 3.21 (12) | 4.85 (8) | 3.59 (24) | 4.12 (14) | 4.87 (26)
  Cycle 1 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 9 | 0 | 0
  Cycle 1 Day 15 |  |  |  |  | 3.47 (19) |  |
  Cycle 1 Day 22: number analyzed (Participants) | 3 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 1 Day 22 | 6.11 (10) |  |  |  |  |  |
  Cycle 3 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 4 | 1
  Cycle 3 Day 1 |  |  |  |  |  | 4.84 (60) | NA (NA) — Not analyzed due to insufficient number of participants.

5. Primary Outcome: Pharmacokinetics -Clearance (Cl) of IMC-CS4
Description: Pharmacokinetics -Clearance (Cl) of IMC-CS4.
Time Frame: Predose, 1, 2, 4 and 8 hours post dose of Cycle 1 Day 1, Cycle 1 Day 15, Cycle 1 Day 22 and Cycle 3 Day 1
Population: All enrolled participants who received at least one dose of study drug and have evaluable PK data for Clearance.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour (L/h)
Arm/Group | 2.5 mg/kg of IMC-CS4 QW | 0.3 mg/kg of IMC-CS4 QW | 0.6 mg/kg of IMC-CS4 QW | 1.25 mg/kg of IMC-CS4 QW | 1.25 mg/kg of IMC-CS4 Q2W | 100 mg of IMC-CS4 QW | 150 mg of IMC-CS4 QW
Number analyzed (Participants) | 6 | 3 | 3 | 5 | 10 | 14 | 8
Liter per hour (L/h)
  Cycle 1 Day 1 | 0.0379 (25) | 0.108 (19) | 0.0715 (28) | 0.0561 (30) | 0.0566 (35) | 0.0561 (43) | 0.0534 (34)
  Cycle 1 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 9 | 0 | 0
  Cycle 1 Day 15 |  |  |  |  | 0.0530 (34) |  |
  Cycle 1 Day 22: number analyzed (Participants) | 3 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 1 Day 22 | 0.0195 (40) |  |  |  |  |  |
  Cycle 3 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 4 | 1
  Cycle 3 Day 1 |  |  |  |  |  | 0.0210 (67) | NA (NA) — Not analyzed due to insufficient number of participants.

6. Secondary Outcome: Recommend Phase 2 Dose (RP2D) of IMC-CS4
Description: The recommended Phase 2 dose was the highest dose where less than 1/3 of participants experienced dose limiting toxicities (DLTs). A DLT is defined as an adverse event (AE) occurring during Cycle 1 that fulfilled 1 of the following criteria: Any Common Terminology Criteria for Adverse Events (CTCAE), version (v) 4.0 Grade 4 neutropenia lasting ≥ 7 days, Grade 3 or 4 neutropenia complicated by fever ≥38.0°C or infection, Grade 4 thrombocytopenia, Grade 3 thrombocytopenia complicated by hemorrhage, Grade 3 or 4 anemia, Grade ≥3 AST/ALT elevation, Grade ≥2 AST/ALT elevation and Grade ≥2 bilirubin elevation and Grade 3 or 4 nonhematologic toxicity. A summary of other nonserious AEs and all Serious Adverse Events (SAE), regardless of causality is located in the Reported Adverse Event section.
Time Frame: Cycle 1 (6 Days)
Population: All enrolled participants who received at least 1 dose of study drug.
Measure: Number; unit: milligrams/week
Groups:
- Phase I Participants: Participants received 2.5 mg/kg QW, 0.3 mg/kg QW, 0.6 mg/kg QW, 1.25 mg/kg Q2W and1.25 mg/kg QW of IMC CS4 in Part A and 100 mg QW, 100 mg QW on weeks 1, 2, 4 and 5 in the Expanded Phase, and 150 mg QW of IMC CS4 by intravenous infusion in Part B.
Arm/Group | Phase I Participants
Number analyzed (Participants) | 36
milligrams/week | 100

7. Secondary Outcome: Percentage of Participants With Anti-IMC-CS4 Antibody Assessment
Description: The overall percentage of participants with treatment-emergent positive for anti-IMC-CS4 antibodies during the study. Participants were considered positive for anti-IMC-CS4 antibodies if they exhibited a post-treatment antibody level that exceeded the positive upper cut point determined from the normal anti-IMC-CS4 level seen in healthy untreated individuals.
Time Frame: Up To 6 Months
Population: All enrolled participants who received at least 1 dose of study drug and have baseline and post baseline data for anti-IMC-CS4 antibodies.
Measure: Number; unit: Percentage of Participants
Groups:
- Cohort 1 (2.5 mg/kg QW): Participants received 2.5 milligram per kilogram (mg/kg) of IMC-CS4 once weekly by intravenous infusion.
Arm/Group | Cohort 1 (2.5 mg/kg QW) | Cohort 2 (0.3 mg/kg QW) | Cohort 3 (0.6 mg/kg QW) | Cohort 4 (1.25 mg/kg Q2W) | Cohort 4 Expanded (1.25 mg/kg Q2W) | Cohort 5 (1.25 mg/kg QW) | Cohort 6a (100 mg QW) | Cohort 6a Expanded (100 mg QW) | Cohort 7a (150 mg QW)
Number analyzed (Participants) | 4 | 3 | 3 | 5 | 3 | 4 | 3 | 11 | 9
Percentage of Participants | 50 | 0 | 0 | 0 | 0 | 25 | 0 | 18.2 | 0

ADVERSE EVENTS:
Time Frame: Up To 6 Months
Description: All enrolled participants
Arm/Group | Cohort 1 (2.5 mg/kg QW) | Cohort 2 (0.3 mg/kg QW) | Cohort 3 (0.6 mg/kg QW) | Cohort 4 (1.25 mg/kg Q2W) | Cohort 4 Expanded (1.25 mg/kg Q2W) | Cohort 5 (1.25 mg/kg QW) | Cohort 6a (100 mg QW) | Cohort 6a Expanded (100 mg QW) | Cohort 7a (150 mg QW)
All-Cause Mortality (participants affected / at risk) | 0/6 | 2/4 | 1/3 | 1/6 | 1/5 | 1/5 | 1/3 | 2/11 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/6 | 1/4 | 2/3 | 2/6 | 2/5 | 3/5 | 1/3 | 4/11 | 3/9
Other Adverse Events (participants affected / at risk) | 6/6 | 4/4 | 3/3 | 6/6 | 4/5 | 3/5 | 3/3 | 11/11 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (2.5 mg/kg QW) (N=6) | Cohort 2 (0.3 mg/kg QW) (N=4) | Cohort 3 (0.6 mg/kg QW) (N=3) | Cohort 4 (1.25 mg/kg Q2W) (N=6) | Cohort 4 Expanded (1.25 mg/kg Q2W) (N=5) | Cohort 5 (1.25 mg/kg QW) (N=5) | Cohort 6a (100 mg QW) (N=3) | Cohort 6a Expanded (100 mg QW) (N=11) | Cohort 7a (150 mg QW) (N=9)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal incarcerated hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sudden death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Cohort 1 (2.5 mg/kg QW) (N=6) | Cohort 2 (0.3 mg/kg QW) (N=4) | Cohort 3 (0.6 mg/kg QW) (N=3) | Cohort 4 (1.25 mg/kg Q2W) (N=6) | Cohort 4 Expanded (1.25 mg/kg Q2W) (N=5) | Cohort 5 (1.25 mg/kg QW) (N=5) | Cohort 6a (100 mg QW) (N=3) | Cohort 6a Expanded (100 mg QW) (N=11) | Cohort 7a (150 mg QW) (N=9)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 2 (6) | 1 (1) | 3 (4) | 1 (1) | 2 (11) | 5 (8) | 5 (10)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 1 (3) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrioventricular block (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 2 (2)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (7) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Deafness unilateral (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Eye swelling (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eyelid oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Periorbital oedema (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 2 (3)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 2 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 2 (4) | 2 (3)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (4) | 3 (5) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (2) | 1 (2) | 2 (4) | 2 (3) | 2 (4) | 2 (2) | 3 (4) | 4 (6)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Retching (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Sensitivity of teeth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (2) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 3 (6)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Face oedema (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Facial pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 2 (3) | 3 (5) | 5 (6) | 2 (3) | 1 (1) | 2 (4) | 6 (10) | 5 (9)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Localised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Medical device pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 2 (5) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nail infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 0/3 (0) | 0/1 (0) | 1/2 (1) | 0/1 (0) | 0/4 (0) | 0/2 (0) | 0/2 (0) | 0/7 (0) | 0/3 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 1 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 4 (27) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 4 (9) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 1 (2) | 2 (3) | 7 (9) | 6 (9)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood cholesterol increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatine phosphokinase (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Blood creatine phosphokinase bb increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 4 (10) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 5 (13) | 5 (12)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (5) | 2 (2) | 1 (2)
Blood lactate dehydrogenase increased (Investigations) | 2 (4) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4)
Blood phosphorus (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood phosphorus decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Electrocardiogram qt prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (4) | 2 (5) | 4 (8) | 2 (6)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0) | 2 (3) | 1 (1) | 1 (1) | 0 (0) | 2 (15) | 2 (14) | 2 (4)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Red blood cells urine positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory rate increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Troponin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urine output decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 1 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Weight increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (5) | 0 (0)
White blood cell count decreased (Investigations) | 2 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (11) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 3 (5) | 1 (2) | 1 (1) | 1 (2) | 2 (2) | 1 (1) | 4 (5) | 4 (6)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 1 (6) | 2 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 3 (6) | 2 (2) | 3 (5) | 1 (2) | 2 (3) | 3 (4) | 3 (5)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 4 (6) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (3) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 2 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 2 (4) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 2 (2)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 1 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (4) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac neoplasm unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (3) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (6) | 1 (7)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Monoplegia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nerve root compression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abnormal dreams (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemoglobinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephropathy (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (5) | 2 (2) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 0/3 (0) | 0/1 (0) | 0/2 (0) | 0/1 (0) | 0/4 (0) | 0/2 (0) | 0/2 (0) | 0/7 (0) | 1/3 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0/3 (0) | 0/1 (0) | 0/2 (0) | 0/1 (0) | 0/4 (0) | 0/2 (0) | 1/2 (1) | 1/7 (1) | 0/3 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 3 (4) | 4 (4) | 3 (4)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (5)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Butterfly rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (3) | 0 (0) | 1 (5) | 1 (2) | 1 (1) | 1 (3) | 1 (2) | 2 (2) | 2 (3)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3)
Pallor (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2015-09-03): https://cdn.clinicaltrials.gov/large-docs/58/NCT01346358/Prot_000.pdf
  • Statistical Analysis Plan (2012-10-19): https://cdn.clinicaltrials.gov/large-docs/58/NCT01346358/SAP_001.pdf